CLINICAL TRIAL: NCT04801108
Title: Combined Zephyr Valve System With Inter-lobar Fissure Completion for Lung Volume Reduction in Emphysema: A Pilot Randomized Controlled Trial
Brief Title: Combined Zephyr Valve System With Inter-lobar Fissure Completion for Lung Volume Reduction in Emphysema
Acronym: COMPLETE-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Pulmonx Corporation (Industry)
Responsible Party: Principal Investigator, Adnan Majid, MD, Chief Interventional Pulmonology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000049
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Emphysema or COPD
Keywords: COPD; Endobronchial valves; Emphysema; Video-assisted thoracic surgery; Robotic thoracic surgery
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Robotics

STUDY DESIGN:
Intervention Model Description: This pilot randomized controlled trial is expected to enroll a total of 20 subjects with a follow-up period of 3 months. All interventions and follow-up will be performed at the BIDMC. Patients will be randomized to an intervention or medical management group using an opaque envelope technique in a 2-4 block pattern to assure a random and evenly distributed patient population.
  After the patient allocated to the medical management, the arm is followed for 3 months, they will be offered the robotic or VATS fissure completion procedure. It will be completely up to the candidates to undergo the intervention. If they decide that they want to proceed with surgery, the previously described methods will be used including the same surgical technique, same postoperative management, and same follow-up timelines and datapoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Medical management group (No Intervention): COPD patients with severe emphysema and incomplete lobar fissures will be placed on maximal medical therapy for 3 months. At the end of this 3 month period, patients will fill in an additional set of quality of life questionnaires including the St.George Respiratory Questionnaire, COPD Assessment tool, and the modified medical research council dyspnea scale. New pulmonary function testing will be performed and crossover to the intervention group will be offered.
- Intervention group (Experimental): COPD patients with severe emphysema and incomplete lobar fissures will undergo video-assisted thoracic surgery fissure completion and valves placement. After a 3 month follow-up period, patients will fill additional quality of life questionnaires including the St.George Respiratory Questionnaire, COPD Assessment tool, and the modified medical research council dyspnea scale. Pulmonary function testing and a high-resolution CT scan will be performed at the end of the 3-month postoperative follow-up.
  Interventions: Procedure: Robotic or VATS lobar fissure completion; Device: Endobronchial valves placement
- Crossover group (Experimental): Subjects allocated to the medical management group will be offered to crossover after the 3 months follow-up period. The same procedure as in the intervention group will be performed. Follow-up after surgery will be the same as in the intervention group.
  Interventions: Procedure: Robotic or VATS lobar fissure completion; Device: Endobronchial valves placement

INTERVENTIONS:
Procedure: Robotic or VATS lobar fissure completion — The lobar fissure adjacent to the target lobe will be completed using a surgical stapler through robotic or video-assisted thoracic surgery.
  Arms: Crossover group; Intervention group
Device: Endobronchial valves placement — Endobronchial valves will be placed in the target lobe after the fissure completion.
  Arms: Crossover group; Intervention group

SUMMARY:
The purpose of this protocol is to perform a pilot prospective randomized controlled clinical trial to evaluate the potential role of lung fissure completion strategy (experimental intervention) in addition to endobronchial valve (EBV) placement (representing "standard-of-care") in select patients with severe COPD/emphysema and with evidence for <95% fissure completion between adjacent lung lobes. In select patients, lung fissure completion strategy will be performed by either video-assisted thorascopic surgery (VATS)-guided or robotic-guided stapling along the lung fissures in an attempt to reduce collateral ventilation and determine whether or not this experimental strategy will improve outcome following subsequent EBV placement. EBV placement will follow successful VATS-guided or robotic-guided fissure stapling.

The study will enroll approximately 20 patients at BIDMC, and outcomes will focus on procedure-related complications, physiological measurements (ex., FEV1 by pulmonary function testing) and clinical symptoms (i.e., questionnaires). Patient will be followed for 3-month period, receiving usual standard of care during the 3 months of follow-up. The goal of this protocol is to determine if elimination of significant collateral lung ventilation between lung lobes is possible, and whether such strategy to eliminate collateral lung ventilation between lobes improves outcomes following subsequent EBV placement (i.e. promotes atelectasis of diseased lung segments) in the management of severe COPD/emphysema in appropriate candidates. For subjects in the medical management control group, upon completion of the 3-month F/U period, they will be eligible for EBV if they choose.

DETAILED DESCRIPTION:
We plan to approach all EBVs candidates that have < 95% lobar fissure completion. Once the patient agrees to participate and sign the consent, all the screening information collected as part of the standard of care will be extracted retrospectively from the medical records including appointment details, 6MWD, and PFTs results. In addition, during the same visit, health-related quality of life will be measured using the Saint George Respiratory Questionnaire (SGRQ) and COPD Assessment Test (CAT), and dyspnea will be assessed with the self-reported modified Medical Research Council dyspnea scale (mMRC). After completing these questionnaires and indexes, subjects will be randomized by an opaque envelope technique following a block 2-4 pattern to either Group 1 (Combined robotic or VATS-fissure completion and BLVR with EBVs) or Group 2 (Medical management).

Both surgical stapling for fissure completion and EBVs implantation will be performed during the same procedure and under general anesthesia in the operating room. Depending on the duration of the surgical intervention, the endoscopic valve implantation might be deferred and performed within 48 hours, based on the clinical judgment of the PI, surgeon, and anesthesiologist present during the procedure.

Initial Bronchoscopic Evaluation Initial flexible bronchoscopy will be done by the interventional pulmonologist who will perform the endoscopic valve placement as part of the standard of care. The bronchoscope will be passed via the endotracheal tube and the major airways will be examined. A bronchial wash will be performed with samples sent for culture. If there are unexpected findings, such as a lesion suspicious for carcinoma or secretions suggesting infection, then appropriate clinical samples will be obtained, and the subject will be re-evaluated to determine if they are eligible to undergo the study procedure later. If so, the procedure will be rescheduled. If not, the subject will be withdrawn from the study and will be considered as an "Enrollment Failure" and recorded as such for statistical analysis.

First Chartis Pulmonary System Evaluation of CV Following initial bronchoscopy, evaluation of CV using the Chartis system (Pulmonx Inc., Redwood, CA, USA), will be performed also as part of the standard of care of the patients. If there is no evidence of CV between the target lobe and the adjacent one, the patient will be withdrawn from the study and EBVs will be placed. On the other hand, if the ChartisTM evaluation is positive for CV, the bronchoscope will be withdrawn, and the patient will undergo robotic or VATS completion of the inter-lobar fissure adjacent to the previously selected target lobe.

Robotic or VATS Inter-Lobar Fissure Completion Surgery will be performed with a robotic or VATS approach under inhaled anesthetic agents by an experienced thoracic surgeon from BIDMC. A double-lumen endotracheal tube will be inserted allowing one-lung ventilation and the maximal collapse of the operative lung. The subject will be placed in lateral decubitus with the operative side up. Through small incisions, the surgeon will create a camera port through the intercostal space and then the anterior and posterior inferior ports. Electrocautery will be used for dissection and exposure of the anterior aspect of the hilum. Stapling will then be performed on the incomplete fissure adjacent to the target lobe, using the Endo GIATM (CovidienTM, Mansfield, MA).

An attempt at conversion to a complete fissure will be made, though depending on the anatomy, it may be possible that residual incomplete fissure of up to 5% may be tolerated. Hemostasis will be evaluated. Sterile water will then be used to fill the surgical area, followed by lung inflation and inspection to verify for air leaks at the level of the stapling. If an air leak is detected, suturing, re-stapling, or applying pleural sealants will be used to seal it. If the air leak persists at the site of stapling despite these measures, the subject will still be allowed to proceed to EBVs implantation. Once the fissure is surgically completed, a chest tube will be installed and connected to a digital chest drainage system (ThopazTM Digital Chest Drainage System, Medela Healthcare).

Second Chartis Pulmonary System Evaluation of CV The double-lumen endotracheal tube will be removed, and a single-lumen tube (8.0 to 8.5 mm) inserted. The lung will be completely re-inflated before this evaluation to return them to normal anatomy. Assessment of CV with the ChartisTM system will be performed once again in the same inter-lobar fissure as before following the previously described methods. If the result is negative for CV or there is an improvement in the evaluation, then we will proceed with EBVs implantation.

EBVs Placement Bronchoscopic placement of EBVs will then be performed as part of the standard of care of patients since they meet the previously mentioned inclusion criteria and have no CV, same as patients with an initial negative ChartisTM evaluation. The airway sizing system and a calibrated balloon will be used in the previous re-inflated lung to determine the appropriate Zephyr® valves size to treat the target lobe airways. The treatment algorithm is complete occlusion of one lobe by using valves to occlude all segments of the lobe. Either upper or lower lobes may be targeted for treatment. The lobe will have been selected by the CT core laboratory based on imaging with computed tomography. However, the PI can choose the alternate eligible lobe if the airway in the primary eligible lobe is overly challenging for valve implantation, such as difficulty associated with the underlying airway anatomy.

A valve may be removed and replaced with a different size valve during the procedure and a valve may also be removed and replaced to improve the location. However, a valve may not be repositioned during the procedure. It is intended that the investigator occlude all segments of the target lobe by placing valves into segmental or sub-segmental airways. There is anatomic variability in the number and size of segments in a lobe, so this protocol does not have a limit on the number of valves to be used. Subjects who do not have any endobronchial valves placed at the end of the bronchoscopy procedure will be withdrawn.

Follow-up Period After BLVR with EBVs, patients will be placed on a standardized follow-up protocol used for individuals that underwent BLVR. All procedures and appointments following EBV placement will be considered standard of care. Data from follow-up appointments at 14 days and 3 months will be collected from the medical records retrospectively including appointment details, complications, CT-scan results, 6MWD, and PFTs results. TLVR will be assessed at 3 months using the CT scans performed on patients as part of their standard of care. The only procedures that will be considered research after the initial surgical intervention would be the measurement of health-related quality of life with the SGRQ and CAT, and dyspnea assessment with the self-reported mMRC at every follow-up appointment.

Crossover Group After the patient allocated to the medical management, the arm is followed for 3 months, they will be offered the robotic or VATS fissure completion procedure. It will be completely up to the candidates to undergo the intervention. If they decide that they want to proceed with surgery, the previously described methods will be used including the same surgical technique, same postoperative management, and same follow-up timelines and datapoints.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years.
* Stable with less than 10mg prednisone (or equivalent) daily.
* Nonsmoking for 4 months prior to screening and willing to not smoke during the study duration.
* Completed a supervised pulmonary rehabilitation program less than equal to 12 months prior to the baseline exam or is regularly performing maintenance respiratory rehabilitation if initial supervised therapy occurred greater than 12 months prior.
* Current pneumococcus vaccination.
* Current influenza vaccination.
* Willing and able to complete protocol required study follow-up assessments and procedures.

Exclusion Criteria:

* > 95% fissure completion on high-resolution chest CT-scan (HRCT) or StratX evaluation with a Chartis evaluation negative for collateral ventilation.
* Clinically significant (greater than 4 tablespoons per day) mucus production.
* Myocardial infarction within 6 months of screening.
* Uncontrolled congestive heart failure.
* Three or more pneumonia episodes in last year.
* Three or more COPD exacerbation episodes in the last year.
* Prior lung transplant, LVRS, bullectomy, or lobectomy.
* Clinically significant bronchiectasis.
* Unable to safely discontinue anticoagulants or platelet activity inhibitors for 7 days.
* Uncontrolled pulmonary hypertension (systolic pulmonary arterial pressure >45mmHg) or evidence or history of CorPulmonale as determined by a recent echocardiogram (completed within the last 3 months prior to screening visit).
* Left ventricular ejection fraction (LVEF) less than 40% as determined by a recent echocardiogram (completed within the last 3 months prior to screening visit).
* Resting bradycardia (<50 beats/min), frequent multifocal PVCs, complex ventricular arrhythmia, sustained SVT.
* Post-bronchodilator FEV1 less than 15% or greater than 45% of the predicted value at screening.
* TLC less than 100% predicted (determined by body plethysmography at screening).
* RV less than 150% predicted in patients with heterogeneous emphysema or less than 200% predicted in patients with homogeneous emphysema (determined by body plethysmography at screening).
* DLCO less than 20% of the predicted value at screening.
* Post-rehabilitation 6-minute walk distance less than 100 meters or greater than 450 meters at screening.
* PaCO2 greater than 50mmHg on room air at screening.
* PaO2 less than 45mmHg on room air at screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Prove that inter-lobar fissures can be completed to at least 95% via robotic thoracic surgery or VATS in severe emphysema patients | 2 years
  We will determine that we met this feasibility objective if the target inter-lobar fissure can be completed in at least 90% of the patients undergoing surgery.
Prove that patients consented for the procedure will ultimately undergo the intervention | 2 years
  We will determine that the study is feasible if at least 90% of consented patients in the intervention arm undergo the procedure.
Incidence of severe adverse events | Through study completion, an average of 2 years
  We will actively monitor and record the severe adverse events that require any kind of additional intervention (medical or surgical) during and after the combined procedure. In case the treating physicians consider that the complications seen in patients outweigh the benefits obtained, the surgical technique will be revised and possible changes will be discussed.

SECONDARY OUTCOMES:
Percentage of patients to achieve target lung volume reduction | 2 years
  Describe the percentage of patients that achieve target lung volume reduction of at least 350mL at three months after the combined procedure.
Percentage of patients with quality of life improvement | 2 years
  Describe the changes in quality of life based on three subjective questionnaires that will be given to patients at baseline and three months after any intervention.
Percentage of patients with significant changes in pulmonary function testing | 2 years
  Describe the changes in PFTs after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheaton AG, Cunningham TJ, Ford ES, Croft JB; Centers for Disease Control and Prevention (CDC). Employment and activity limitations among adults with chronic obstructive pulmonary disease--United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 Mar 27;64(11):289-95. PMID 25811677
- [Background] "Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary." Claus F. Vogelmeier, Gerard J. Criner, Fernando J. Martinez, Antonio Anzueto, Peter J. Barnes, Jean Bourbeau, Bartolome R. Celli, Rongchang Chen, Marc Decramer, Leonardo M. Fabbri, Peter Frith, David M.G. Halpin, M. Victorina Lopez Varela, Masaharu Nishimura, Nicolas Roche, Roberto Rodriguez-Roisin, Don D. Sin, Dave Singh, Robert Stockley, Jorgen Vestbo, Jadwiga A. Wedzicha and Alvar Agusti. Eur Respir J 2017; 49: 1700214. Eur Respir J. 2017 Jun 22;49(6):1750214. doi: 10.1183/13993003.50214-2017. Print 2017 Jun. No abstract available. PMID 28642306
- [Background] Hartman JE, Vanfleteren LEGW, van Rikxoort EM, Klooster K, Slebos DJ. Endobronchial valves for severe emphysema. Eur Respir Rev. 2019 Apr 17;28(152):180121. doi: 10.1183/16000617.0121-2018. Print 2019 Jun 30. PMID 30996040
- [Background] Majid A, Kheir F, Alape D, Chee A, Parikh M, DeVore L, Agnew A, Gangadharan S. Combined Thoracoscopic Surgical Stapling and Endobronchial Valve Placement For Lung Volume Reduction With Incomplete Lobar Fissures: An Experimental Pilot Animal Study. J Bronchology Interv Pulmonol. 2020 Apr;27(2):128-134. doi: 10.1097/LBR.0000000000000617. PMID 31436607
- [Background] Celli BR, Wedzicha JA. Update on Clinical Aspects of Chronic Obstructive Pulmonary Disease. N Engl J Med. 2019 Sep 26;381(13):1257-1266. doi: 10.1056/NEJMra1900500. No abstract available. PMID 31553837
- [Background] Kochanek KD, Murphy S, Xu J, Arias E. Mortality in the United States, 2016. NCHS Data Brief. 2017 Dec;(293):1-8. PMID 29319473
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Sullivan SD, Ramsey SD, Lee TA. The economic burden of COPD. Chest. 2000 Feb;117(2 Suppl):5S-9S. doi: 10.1378/chest.117.2_suppl.5s. PMID 10673466
- [Background] Rennard SI. COPD: overview of definitions, epidemiology, and factors influencing its development. Chest. 1998 Apr;113(4 Suppl):235S-241S. doi: 10.1378/chest.113.4_supplement.235s. PMID 9552012
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Maltais F. Exercise and COPD: therapeutic responses, disease-related outcomes, and activity-promotion strategies. Phys Sportsmed. 2013 Feb;41(1):66-80. doi: 10.3810/psm.2013.02.2001. PMID 23445862
- [Background] Fishman A, Martinez F, Naunheim K, Piantadosi S, Wise R, Ries A, Weinmann G, Wood DE; National Emphysema Treatment Trial Research Group. A randomized trial comparing lung-volume-reduction surgery with medical therapy for severe emphysema. N Engl J Med. 2003 May 22;348(21):2059-73. doi: 10.1056/NEJMoa030287. Epub 2003 May 20. PMID 12759479
- [Background] Fessler HE, Permutt S. Lung volume reduction surgery and airflow limitation. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):715-22. doi: 10.1164/ajrccm.157.3.9608004. PMID 9517581
- [Background] Naunheim KS, Wood DE, Krasna MJ, DeCamp MM Jr, Ginsburg ME, McKenna RJ Jr, Criner GJ, Hoffman EA, Sternberg AL, Deschamps C; National Emphysema Treatment Trial Research Group. Predictors of operative mortality and cardiopulmonary morbidity in the National Emphysema Treatment Trial. J Thorac Cardiovasc Surg. 2006 Jan;131(1):43-53. doi: 10.1016/j.jtcvs.2005.09.006. Epub 2005 Dec 5. PMID 16399293
- [Background] DeCamp MM Jr, McKenna RJ Jr, Deschamps CC, Krasna MJ. Lung volume reduction surgery: technique, operative mortality, and morbidity. Proc Am Thorac Soc. 2008 May 1;5(4):442-6. doi: 10.1513/pats.200803-023ET. PMID 18453353
- [Background] DeCamp MM, Blackstone EH, Naunheim KS, Krasna MJ, Wood DE, Meli YM, McKenna RJ Jr; NETT Research Group. Patient and surgical factors influencing air leak after lung volume reduction surgery: lessons learned from the National Emphysema Treatment Trial. Ann Thorac Surg. 2006 Jul;82(1):197-206; discussion 206-7. doi: 10.1016/j.athoracsur.2006.02.050. PMID 16798215
- [Background] Labarca G, Uribe JP, Pacheco C, Folch E, Kheir F, Majid A, Jantz MA, Mehta HJ, Patel N, Herth FJF, Fernandez-Bussy S. Bronchoscopic Lung Volume Reduction with Endobronchial Zephyr Valves for Severe Emphysema: A Systematic Review and Meta-Analysis. Respiration. 2019;98(3):268-278. doi: 10.1159/000499508. Epub 2019 May 22. PMID 31117102
- [Background] Sciurba FC, Ernst A, Herth FJ, Strange C, Criner GJ, Marquette CH, Kovitz KL, Chiacchierini RP, Goldin J, McLennan G; VENT Study Research Group. A randomized study of endobronchial valves for advanced emphysema. N Engl J Med. 2010 Sep 23;363(13):1233-44. doi: 10.1056/NEJMoa0900928. PMID 20860505
- [Background] Eberhardt R, Gompelmann D, Schuhmann M, Reinhardt H, Ernst A, Heussel CP, Herth FJF. Complete unilateral vs partial bilateral endoscopic lung volume reduction in patients with bilateral lung emphysema. Chest. 2012 Oct;142(4):900-908. doi: 10.1378/chest.11-2886. PMID 22459779
- [Background] Shah PL, Herth FJ. Current status of bronchoscopic lung volume reduction with endobronchial valves. Thorax. 2014 Mar;69(3):280-6. doi: 10.1136/thoraxjnl-2013-203743. Epub 2013 Sep 5. PMID 24008689
- [Background] Cetti EJ, Moore AJ, Geddes DM. Collateral ventilation. Thorax. 2006 May;61(5):371-3. doi: 10.1136/thx.2006.060509. PMID 16648350
- [Background] Koster TD, Slebos DJ. The fissure: interlobar collateral ventilation and implications for endoscopic therapy in emphysema. Int J Chron Obstruct Pulmon Dis. 2016 Apr 13;11:765-73. doi: 10.2147/COPD.S103807. eCollection 2016. PMID 27110109
- [Background] Koster TD, van Rikxoort EM, Huebner RH, Doellinger F, Klooster K, Charbonnier JP, Radhakrishnan S, Herth FJ, Slebos DJ. Predicting Lung Volume Reduction after Endobronchial Valve Therapy Is Maximized Using a Combination of Diagnostic Tools. Respiration. 2016;92(3):150-7. doi: 10.1159/000448849. Epub 2016 Aug 31. PMID 27577190
- [Background] Gompelmann D, Eberhardt R, Slebos DJ, Brown MS, Abtin F, Kim HJ, Holmes-Higgin D, Radhakrishnan S, Herth FJ, Goldin J. Diagnostic performance comparison of the Chartis System and high-resolution computerized tomography fissure analysis for planning endoscopic lung volume reduction. Respirology. 2014 May;19(4):524-30. doi: 10.1111/resp.12253. Epub 2014 Feb 25. PMID 24612306
- [Background] Herth FJ, Eberhardt R, Gompelmann D, Ficker JH, Wagner M, Ek L, Schmidt B, Slebos DJ. Radiological and clinical outcomes of using Chartis to plan endobronchial valve treatment. Eur Respir J. 2013 Feb;41(2):302-8. doi: 10.1183/09031936.00015312. Epub 2012 May 3. PMID 22556025
- [Background] Herth FJF, Slebos DJ, Criner GJ, Valipour A, Sciurba F, Shah PL. Endoscopic Lung Volume Reduction: An Expert Panel Recommendation - Update 2019. Respiration. 2019;97(6):548-557. doi: 10.1159/000496122. Epub 2019 Mar 5. PMID 30836374
- [Background] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Background] Slebos DJ, Shah PL, Herth FJ, Valipour A. Endobronchial Valves for Endoscopic Lung Volume Reduction: Best Practice Recommendations from Expert Panel on Endoscopic Lung Volume Reduction. Respiration. 2017;93(2):138-150. doi: 10.1159/000453588. Epub 2016 Dec 20. PMID 27992862